CLINICAL TRIAL: NCT06125223
Title: A Single-arm, Prospective, Phase II Study of PABLIXIMAB Combined With TP Chemotherapy as Neoadjuvant Therapy for Locally Advanced Head and Neck Squamous-cell Carcinoma
Brief Title: PABLIXIMAB as Neoadjuvant Therapy for Head and Neck Squamous-cell Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Shi Li，MD, Associate Professor, Xijing Hospital
Other Study IDs: KY20232325
Record Dates: First submitted 2023-10-31; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Neoadjuvant Therapy; Immunotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this clinical trial is to learn about the efficacy and safety of pablizumab combined with neoadjuvant chemotherapy in patients with locally advanced head and neck squamous cell carcinoma.

The main question it aims to answer is: Pathological complete remission (PCR) rate of tumor after neoadjuvant immunotherapy.

Participants will be asked to perform CT and MRI of head and neck, ultrasonography of cervical lymph nodes and necessary laboratory examinations Before and after neoadjuvant therapy. And will be following-up for at least 1 year.

DETAILED DESCRIPTION:
The secondary questions it aims to answer are:

Objective response rate (ORR) after neoadjuvant therapy

* R0 resection rate
* major pathological remission (MPR) rate
* organ preservation rate
* event-free survival (EFS)
* local recurrence-free survival (LRFS)
* distant metastasis-free survival (DMFS)
* quality of life score (QoL)
* overall survival (OS)
* incidence of adverse events (including neoadjuvant stage AEs and full course AEs) The exploratory question it aims to answer is: clearance of peripheral blood ctDNA.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-80 years old, including 18 years old and 80 years old;
2. MRI diagnosis of resectable stage III-IVA oropharynx, larynx and hypopharynx squamous-cell carcinoma confirmed by histopathology or cytology;
3. ECOG PS score 0-1;
4. the expression of PD-L1 was detected by immunohistochemistry (TPS and CPS score)
5. having at least one measurable lesion according to RECIST version 1.1;
6. expected survival time ≥6 months;
7. The neutrophil count was ≥1.5 × 10^9/L, the platelet count was ≥100 × 10^9/L, the hemoglobin count was ≥90 g/L
8. renal function was normal: serum creatinine ≤1.5×ULN;
9. the liver function was basically normal: serum total bilirubin ≤1.5 × ULN, serum aspartate transaminase (AST)≤2.5×ULN, serum Alanine transaminase (ALT)≤2.5 ×ULN;
10. female patients had to be negative for a urine pregnancy test before the start of the study (not applicable to patients with bilateral oophorectomy and/or hysterectomy or postmenopausal patients) ;
11. Sign the written informed consent.

Exclusion Criteria:

1. patients were treated with anti-tumor drugs including but not limited to PD-1 inhibitor, CTLA-4 antibody, EGFR monoclonal antibody, EGFR-tki, and anti-angiogenesis drugs;
2. History of autoimmune diseases including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, Rheumatoid Arthritis, inflammatory bowel disease, Antiphospholipid syndrome vascular thrombosis, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis or glomerulonephritis.
3. participated in other intervention clinical trials within 30 days before screening;
4. history of other malignancies (except cured skin basal-cell carcinoma) ;
5. the presence of serious and poorly controlled co-morbidities (e.g. heart failure, diabetes, hypertension, liver failure, kidney failure, thyroid disease, mental illness, etc.) ;
6. Known to be infected with HIV or active hepatitis or tuberculosis;
7. major surgery or planned surgery within 30 days before the first dose of the trial drug;
8. Persons who are allergic to the use of drugs or their components in the programme;
9. pregnancy (confirmed by blood or urine HCG testing) or lactation in women, or in subjects of reproductive age who were unwilling or unable to use effective contraception (for both male and female subjects) until at least 6 months after the last trial treatment;
10. it is not suitable for the researcher to participate in this study;
11. Unwilling to participate in the study or unable to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A otolaryngology patient at Xijing Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission (pCR) rate of tumor after neoadjuvant immunotherapy. | About 50 days after the start of neoadjuvant immunotherapy.
  pCR means that there are no residual living tumor cells in the tumor bed and lymph nodes after neoadjuvant therapy.

SECONDARY OUTCOMES:
ORR(objective response rate) | At least 1 year.
  Objective response rates after neoadjuvant immunotherapy were measured, usually as the proportion of patients whose tumor volume decreased by 30% and maintained over 4 weeks, that is, the sum of the rates of complete response (CR) and partial response (PR) , the higher the ORR, the more patients achieved tumor shrinkage with the treatment.
R0 resection rate | At least 1 year.
  R0 resection is the highest standard of tumor resection, which means complete tumor resection with negative margin. The tumor R0 resection rate was calculated for the patients who underwent surgery after the completion of neoadjuvant immunotherapy.
MPR（major pathological response） | At least 1 year.
  MPR is defined as the percentage of residual tumor cells in the tumor bed being less than or equal to 10% .
Overall survival rate | At least 1 year.
  Overall survival is the proportion of all participants who survived the study period. Overall survival was calculated by dividing the number of people alive by the total number at the start of the study.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | At least 1 year.
  Researchers should grade the severity of each adverse event. If the severity/intensity of an adverse event is not specified in the guidelines, the investigator can assess it based on the general definition of grade 1-5 and in conjunction with his or her medical judgment.

OTHER OUTCOMES:
clearance of peripheral blood ctDNA | At least 1 year.
  ctDNA is circulating tumor DNA, also known as tumor DNA, which enters the bloodstream when tumor cells die or are released. It is a liquid biopsy method that detects the presence and associated changes of tumor cells in a blood sample.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Johnson DE, Burtness B, Leemans CR, Lui VWY, Bauman JE, Grandis JR. Head and neck squamous cell carcinoma. Nat Rev Dis Primers. 2020 Nov 26;6(1):92. doi: 10.1038/s41572-020-00224-3. PMID 33243986
- [Result] Keam B, Machiels JP, Kim HR, Licitra L, Golusinski W, Gregoire V, Lee YG, Belka C, Guo Y, Rajappa SJ, Tahara M, Azrif M, Ang MK, Yang MH, Wang CH, Ng QS, Wan Zamaniah WI, Kiyota N, Babu S, Yang K, Curigliano G, Peters S, Kim TW, Yoshino T, Pentheroudakis G. Pan-Asian adaptation of the EHNS-ESMO-ESTRO Clinical Practice Guidelines for the diagnosis, treatment and follow-up of patients with squamous cell carcinoma of the head and neck. ESMO Open. 2021 Dec;6(6):100309. doi: 10.1016/j.esmoop.2021.100309. Epub 2021 Nov 26. PMID 34844180
- [Result] Caudell JJ, Gillison ML, Maghami E, Spencer S, Pfister DG, Adkins D, Birkeland AC, Brizel DM, Busse PM, Cmelak AJ, Colevas AD, Eisele DW, Galloway T, Geiger JL, Haddad RI, Hicks WL, Hitchcock YJ, Jimeno A, Leizman D, Mell LK, Mittal BB, Pinto HA, Rocco JW, Rodriguez CP, Savvides PS, Schwartz D, Shah JP, Sher D, St John M, Weber RS, Weinstein G, Worden F, Yang Bruce J, Yom SS, Zhen W, Burns JL, Darlow SD. NCCN Guidelines(R) Insights: Head and Neck Cancers, Version 1.2022. J Natl Compr Canc Netw. 2022 Mar;20(3):224-234. doi: 10.6004/jnccn.2022.0016. PMID 35276673
- [Result] Bhatia A, Burtness B. Treating Head and Neck Cancer in the Age of Immunotherapy: A 2023 Update. Drugs. 2023 Feb;83(3):217-248. doi: 10.1007/s40265-023-01835-2. Epub 2023 Jan 16. PMID 36645621
- [Result] Veigas F, Mahmoud YD, Merlo J, Rinflerch A, Rabinovich GA, Girotti MR. Immune Checkpoints Pathways in Head and Neck Squamous Cell Carcinoma. Cancers (Basel). 2021 Mar 1;13(5):1018. doi: 10.3390/cancers13051018. PMID 33804419
- [Result] Hamid O, Robert C, Daud A, Hodi FS, Hwu WJ, Kefford R, Wolchok JD, Hersey P, Joseph R, Weber JS, Dronca R, Mitchell TC, Patnaik A, Zarour HM, Joshua AM, Zhao Q, Jensen E, Ahsan S, Ibrahim N, Ribas A. Five-year survival outcomes for patients with advanced melanoma treated with pembrolizumab in KEYNOTE-001. Ann Oncol. 2019 Apr 1;30(4):582-588. doi: 10.1093/annonc/mdz011. PMID 30715153
- [Result] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Result] Diaz LA Jr, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fourchardiere C, Rivera F, Elez E, Le DT, Yoshino T, Zhong WY, Fogelman D, Marinello P, Andre T; KEYNOTE-177 Investigators. Pembrolizumab versus chemotherapy for microsatellite instability-high or mismatch repair-deficient metastatic colorectal cancer (KEYNOTE-177): final analysis of a randomised, open-label, phase 3 study. Lancet Oncol. 2022 May;23(5):659-670. doi: 10.1016/S1470-2045(22)00197-8. Epub 2022 Apr 12. PMID 35427471
- [Result] Oliva M, Spreafico A, Taberna M, Alemany L, Coburn B, Mesia R, Siu LL. Immune biomarkers of response to immune-checkpoint inhibitors in head and neck squamous cell carcinoma. Ann Oncol. 2019 Jan 1;30(1):57-67. doi: 10.1093/annonc/mdy507. PMID 30462163
- [Result] Uppaluri R, Campbell KM, Egloff AM, Zolkind P, Skidmore ZL, Nussenbaum B, Paniello RC, Rich JT, Jackson R, Pipkorn P, Michel LS, Ley J, Oppelt P, Dunn GP, Barnell EK, Spies NC, Lin T, Li T, Mulder DT, Hanna Y, Cirlan I, Pugh TJ, Mudianto T, Riley R, Zhou L, Jo VY, Stachler MD, Hanna GJ, Kass J, Haddad R, Schoenfeld JD, Gjini E, Lako A, Thorstad W, Gay HA, Daly M, Rodig SJ, Hagemann IS, Kallogjeri D, Piccirillo JF, Chernock RD, Griffith M, Griffith OL, Adkins DR. Neoadjuvant and Adjuvant Pembrolizumab in Resectable Locally Advanced, Human Papillomavirus-Unrelated Head and Neck Cancer: A Multicenter, Phase II Trial. Clin Cancer Res. 2020 Oct 1;26(19):5140-5152. doi: 10.1158/1078-0432.CCR-20-1695. Epub 2020 Jul 14. PMID 32665297
- [Result] Ferris RL, Spanos WC, Leidner R, Goncalves A, Martens UM, Kyi C, Sharfman W, Chung CH, Devriese LA, Gauthier H, Chiosea SI, Vujanovic L, Taube JM, Stein JE, Li J, Li B, Chen T, Barrows A, Topalian SL. Neoadjuvant nivolumab for patients with resectable HPV-positive and HPV-negative squamous cell carcinomas of the head and neck in the CheckMate 358 trial. J Immunother Cancer. 2021 Jun;9(6):e002568. doi: 10.1136/jitc-2021-002568. PMID 34083421